CLINICAL TRIAL: NCT02257320
Title: A Feasibility Study of the Bruxoff™ Device to Assess EMG Activity in Subjects Diagnosed With Sleep Bruxism Using TMJ NextGeneration(TM)
Brief Title: TMJ NextGeneration(TM) Feasibility Study
Acronym: Bruxoff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TMJ Health (Industry)
Collaborators: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Organization: Cardiox Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMJ-1002
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feasibility (Other): Assessing EMG activity with Bruxoff(TM) device
  Interventions: Device: TMJ NextGeneration(TM)

INTERVENTIONS:
Device: TMJ NextGeneration(TM) — The TMJ NextGeneration(TM) device consists of a pair of small, hollow ear inserts. These ear inserts are custom-fit to each subject's ear canals. The devices rest in the outer third of the ear canal and have a small retraction post that allows for removal of the device from the ear. The devices conform to the shape of the ear canal when the jaw is in the open position and permit full passage of sound into each ear. The mechanisms of action of the inserts are to support the TMJ and associated secondary musculature to reduce strain in the TMJ area and to provide cognitive awareness to the wearer regarding para-functional habits, i.e., jaw clenching.

SUMMARY:
The study is an open-label, prospective, single-center, non-randomized feasibility study of the Bruxoff(TM) device to identify EMG activity associated with bruxism, and to assess the impact of the TMJ NextGeneration(TM) device upon the occurrence of night-time bruxism events and incidence of migraines and headache in subjects diagnosed with sleep bruxism.

DETAILED DESCRIPTION:
The study will be conducted at one study center in the U.S. Subjects will be enrolled in the trial for a period of 8 weeks. The study will consist of a screening phase lasting up to 2 weeks and a follow up treatment period lasting 8 weeks. Subjects will visit the dental clinic twice during the screening period, then five times during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at least 18 years of age;
2. Subject has had a diagnosis of sleep bruxism;
3. Subject has been medically screened and diagnosed by a physician as having headaches and/or migraines;
4. Subject is willing to comply with the usage instructions for the Bruxoff device;
5. Is able to read and understand the ICF and has voluntarily provided written informed consent.
6. Subject is able to open their mouth at least 17 mm to be fitted for the TMJ NextGenerationTM device;
7. Male Subjects are willing to have a clean shaven face on the nights that the Bruxoff device will be used;
8. Subject agrees that when using the Bruxoff device to keep their cellular phone in another room.

Exclusion Criteria:

1. Subjects with any physical or behavioral disorder, which, in the opinion of the Principal Investigator, may interfere with the use of the device or compliance with the study protocol;
2. Subject has any sleep disorder other than bruxism;
3. Subjects who have had direct trauma to the jaw;
4. Subjects who have had prior TMJ or ear surgery;
5. Subjects who have a narrow ear canal or impression of the ear canal, which is prolapsed due to an anatomical shift or failure of the ear canal wall structure, or a canal that does not allow for the ear canal second turn to be identified;
6. Subjects with visible or congenital ear deformity as observed on targeted physical exam;
7. Subjects whose ear canal anatomy does not allow for fit of the study device;
8. Subjects who have a history of ear pain unrelated to TMJ;
9. Subjects who have a history of ear drainage in the past 6 months;
10. Subjects who have active ear drainage, swelling, or redness as observed on targeted physical exam;
11. Subject has experienced chronic pain (not including migraine pain) associated with sleep bruxism or TMD for more than six months;
12. Subject has a pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Bruxoff(TM) to measure EMG activity in bruxing subjects using the TMJ NextGeneration(TM) device. | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: simon blackburn, Study Director — Cardiox Corporation
Locations (2):
- United States (2):
  - Ear, Nose and Throat Associates of South Florida, Boca Raton, Florida
  - Ear, Nose and Throat Associates of South Florida, Boynton Beach, Florida